CLINICAL TRIAL: NCT02980224
Title: A Randomized, Multicenter, Double-Masked, Placebo-Controlled Study of the Safety and Efficacy of OmegaD Softgels in the Treatment of Dry Eye Disease
Brief Title: Study of the Safety and Efficacy of OmegaD Softgels in the Treatment of Dry Eye Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: OmegaD LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OmegaD-2016-001
Record Dates: First submitted 2016-11-30; First posted 2016-12-02 (Estimated); Results first posted 2019-09-11 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-11

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OmegaD (Experimental): OmegaD Softgels
  Interventions: Drug: OmegaD
- Placebo (Placebo Comparator): Placebo Softgels
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OmegaD — OmegaD Softgels
  Arms: OmegaD
Drug: Placebo — Placebo Softgels
  Arms: Placebo

SUMMARY:
This is a phase 3 study to evaluate the safety and efficacy of OmegaD softgels for the treatment of dry eye disease. A daily dose of 2 OmegaD softgels dosed orally BID will be compared to 2 placebo softgels dosed orally BID for 84 days. Approximately 164 subjects will be evaluated for their signs and symptoms of dry eye disease and for safety throughout the study.

DETAILED DESCRIPTION:
Inflammation is a key component of dry eye disease. Increasing the systemic levels of omega-3 fatty acids relative to omega-6 levels can mediate immune responses. Evaluating whether omega-3 supplementation can improve dry eye disease signs, symptoms and associated measures of inflammation may present a new therapeutic option for dry eye disease.

The primary objective of this study is to evaluate the safety and efficacy of twice daily (BID) dosing of OmegaD softgels in subjects with dry eye disease.

Male and female subjects between 18 years and 90 years of age, with patient-reported dry eye symptoms and a clinical diagnosis of dry eye disease supported by global clinical assessment will be screened and enrolled. Each subject must have, in at least one eye, tear osmolarity of ≥ 312 mOsm/L and meibomian gland dysfunction as defined by a grade of 1 or 2 on the meibomian orifice size scale at both Screening and Baseline in at least one eye. In addition, Tear break up time (TBUT) must be ≤ 7 seconds in both eyes at both Screening and Baseline and the Schirmer's test score in both eye(s) must be ≥ 5 mm at Baseline.

Approximately 164 subjects will be randomized (1:1) to 1 of 2 treatment arms and treated for 84 days (12 weeks) with either OmegaD softgels; 2 softgels BID or placebo softgels; 2 softgels BID. The study will be double-masked with OmegaD and placebo being identical-appearing softgels.

Subjects will participate in safety and efficacy assessments throughout the study. Efficacy assessments will include, tear osmolarity, meibomian gland dysfunction grading, TBUT, Schirmer's Test, and dry eye symptoms based on the OSDI questionnaire, Safety assessments will include, slit lamp examination and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age ≥ 18 years and ≤ 90 years on the date of informed consent.
2. All subjects must provide signed written consent prior to participation in any study related procedures.
3. Patient-reported dry eye symptoms.
4. Clinical diagnosis of dry eye disease supported by global clinical assessment.
5. Presence of tear osmolarity in at least one eye ≥ 312 mOsm/L at both Screening and Baseline.
6. Presence of meibomian gland dysfunction as defined by a grade of 1 or 2 on the meibomian orifice size scale in at least one eye at both Screening and Baseline. The qualifying osmolarity level and meibomian orifice size grade must be present in the same eye at both Screening and Baseline if only one eye qualifies.
7. Female subjects of childbearing potential must have a negative urine pregnancy test at Screening. Women of childbearing potential (i.e., women who are not either postmenopausal for one year or surgically sterile) must use an acceptable form of contraception throughout the study.

Exclusion Criteria:

1. Allergy to fish oil or safflower oil (component of placebo softgels) or any component of the softgel material.
2. Schirmer's test score < 5 mm at Screening in either eye.
3. Tear break-up time > 7 seconds at Screening or Baseline in either eye.
4. Clinically significant eyelid deformity or eyelid movement disorder that is caused by conditions such as notch deformity, incomplete lid closure, entropion, ectropion, hordeolum or chalazion.
5. Active seasonal and/or perennial allergic conjunctivitis or rhinitis.
6. Previous ocular disease leaving sequelae or requiring current topical eye therapy other than for dry eye disease, including, but not limited to: active corneal or conjunctival infection of the eye and ocular surface scarring.
7. History or presence of abnormal nasolacrimal drainage.
8. Laser-assisted in situ keratomileusis (LASIK) or photorefractive keratectomy (PRK) performed within one year prior to Screening and throughout the study period.
9. Ophthalmic drop use within 2 hours prior to any study visit. Any over-the-counter (OTC) artificial tear should be continued at the same frequency and with no change in drop brand.
10. Contact lens wear within 12 hours prior to any study visit; subjects determined to have worn contact lenses within 12 hours must be rescheduled.
11. Punctal cauterization or punctal plug placement within 60 days prior to Screening and throughout the study period.
12. Started or changed the dose of systemic medications known to affect tear production within 30 days prior to Screening and throughout the study period. These include but are not limited to the following medications:

    * Immunomodulators
    * Antihistamines
    * Tricyclic antidepressants
    * Diuretics
    * Corticosteroids (intranasal, inhaled, topical dermatological, and perianal steroids are permitted).
13. Use of any topical prescription ophthalmic medications (including cyclosporine [Restasis®, steroids, nonsteroidal anti-inflammatory drugs [NSAIDs], anti-glaucoma medications), oral tetracyclines or topical macrolides, oral nutraceuticals [fish, flax, black currant seed oils, etc.] within 21 days prior to Screening and throughout the study period.
14. Chronic daily use (defined as > 7 consecutive days at the recommended dosing frequency) of oral NSAIDs during the study period. ANY use of oral NSAIDS during the study period must be discussed with the Medical Monitor.
15. Participation in any drug or device clinical investigation within 30 days prior to entry into this study and/or during the period of study participation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Artesia, California
  - Mission Hills, California
  - Rancho Cordova, California
  - Danbury, Connecticut
  - Crystal River, Florida
  - Deerfield Beach, Florida
  - Fort Myers, Florida
  - Pittsburg, Kansas
  - Edgewood, Kentucky
  - Cincinnati, Ohio
  - Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OmegaD | Placebo
Started | 89 | 91
Completed | 85 | 88
Not Completed | 4 | 3
Not completed — Adverse Event | 4 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OmegaD | Placebo | Total
Number analyzed (Participants) | 89 | 91 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (12.78) | 61.5 (12.53) | 60.6 (12.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 71 | 149
  Male | 11 | 20 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 23 | 52
  Not Hispanic or Latino | 60 | 68 | 128
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 4 | 11
  White | 79 | 82 | 161
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 89 | 91 | 180

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Tear Break up Time(TBUT ) at Day 84
Description: The difference between Baseline (Day 1) and Day 84 in Tear Break Up Time. TBUT is a clinical test used to assess for evaporative dry eye disease. To measure TBUT, fluorescein is instilled into the patient's tear film and the patient is asked not to blink while the tear film is observed under a broad beam of cobalt blue illumination. The TBUT is recorded as the number of seconds that elapse between the last blink and the appearance of the first dry spot in the tear film, as observed via slit lamp examination.
Time Frame: Baseline and 84 Days
Population: Intent to Treat Population
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | OmegaD | Placebo
Number analyzed (Participants) | 89 | 91
seconds | 1.45 (0.261) | 1.23 (0.260)

2. Primary Outcome: Change From Baseline in Dry Eye Symptom Scores (OSDI Questionnaire)
Description: Difference from Baseline (Day 1) to Day 84 in the OSDI Questionnaire (dry eye symptom score). Responses evaluate a subjects experience of a symptom on the following scale:
  0 (none of the time)
  1. (some of the time)
  2. (half of the time)
  3. (most of the time)
  4. (all of the time)
  The 12 questions are as follows:
  Have you experienced any of the following during the last week:
  1. Eyes that are sensitive to light
  2. Eyes that feel gritty
  3. Painful or sore eyes
  4. Blurred vision
  5. Poor vision
     Have problems with your eyes limited you in performance of any of the following during the last week:
  6. Reading
  7. Driving at night
  8. Working with a computer or bank machine (ATM)
  9. Watching TV
     Have your eyes felt uncomfortable in any of the following situations during the last week:
  10. Windy conditions
  11. Places or areas with low humidity (very dry)
  12. Areas that are air conditioned
  A higher score means a worse outcome. The scores for the 12 questions are added together.
Time Frame: Baseline and 84 Days
Population: Intent to Treat Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | OmegaD | Placebo
Number analyzed (Participants) | 89 | 91
score on a scale | -13.39 (1.804) | -15.04 (1.794)

3. Secondary Outcome: The Frequency and Severity of Adverse Events
Description: Number and Percentage of Subjects Reporting Adverse Events
Time Frame: 84 Days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | OmegaD | Placebo
Number analyzed (Participants) | 89 | 91
Participants
  Number of Subjects Reporting AEs | 23 | 16
  Number of Subjects Reporting 0 AEs | 66 | 75
  Number of Subjects Reporting 1 AE | 17 | 9
  Number of Subjects Reporting >1 AE | 6 | 7
  Number of Serious AEs | 0 | 0
  Subjects Reporting AEs leading to Discontinuation | 4 | 1
  Subjects with AEs leading to Drug Interrupti | 1 | 0
  Deaths | 0 | 0

ADVERSE EVENTS:
Time Frame: 84 Days
Arm/Group | OmegaD | Placebo
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/91
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/91
Other Adverse Events (participants affected / at risk) | 12/89 | 1/91
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OmegaD (N=89) | Placebo (N=91)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2016-06-24): https://cdn.clinicaltrials.gov/large-docs/24/NCT02980224/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-06): https://cdn.clinicaltrials.gov/large-docs/24/NCT02980224/SAP_001.pdf